CLINICAL TRIAL: NCT03606720
Title: Effect of Low-level Laser Therapy and Pelvic Stabilisation Exercises on Postpartum Pelvic Girdle Pain
Brief Title: Effect of Low Level Laser Therapy and Pelvic Stabilisation Exercises on Postpartum Pelvic Girdle Pain
Acronym: PGP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, saad shehata, Head of Physical Therapist department in Imbaba general hospital, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 01114933504
Record Dates: First submitted 2018-07-14; First posted 2018-07-31 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Pelvic Girdle Pain
Keywords: Pelvic Girdle Pain; low level laser therapy; pelvic stabilization exercises; postpartum pain
MeSH Terms: conditions — Pelvic Girdle Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: The study were to determine whether the combination of low level laser therapy and pelvic stabilization exercises is more efficient, and possibly effective, treatment protocol in the treatment of pelvic girdle pain,and study and compare the effectiveness of specific stabilizing exercises with low level laser therapy in PGP subjects in terms of pain intensity, functional status and health-related quality of life following delivery
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: If low level laser therapy 810nm and pelvic stabilization exercises can reduce pain and improve function there will be a new treatment option for this condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group(A) low level laser therapy (Experimental): composed of 30 patients who received pelvic stabilization exercises and low level laser therapy For 12 sessions over six week's period by 2 sessions per week.
  Interventions: Other: low level laser therapy; Other: pelvic stabilization exercises
- group(B) pelvic stabilization exercises only (Active Comparator): composed of 30 patients who pelvic stabilization exercises only For 12 sessions over six week's period by 2 sessions per week.
  Interventions: Other: pelvic stabilization exercises
- group (C) low level laser therapy only (Active Comparator): composed of 30 patients who low level laser therapy only For 12 sessions over six week's period by 2 sessions per week.
  Interventions: Other: low level laser therapy

INTERVENTIONS:
Other: low level laser therapy — low level laser therapy (LLLT) is a modality that has been used by the medical profession for decades to treat acute and chronic pain conditions ranging from tendonitis and bursitis, to back pain and pelvic girdle pain.
  Other Names: (LLLT)
  Arms: group (C) low level laser therapy only; group(A) low level laser therapy
Other: pelvic stabilization exercises — special program of pelvic stabilization exercises depending on exercising of transverse abdominal in addition to co activation of lumbar multifidus muscles at the lumbosacral area , exercising of oblique abdominal, gluteus maximus, latissimus dorsi muscles , quadratus lumborum, erector spinae, also, hip abductors and adductors. will done by all patients
  Other Names: (PSE)
  Arms: group(A) low level laser therapy; group(B) pelvic stabilization exercises only

SUMMARY:
This study will be conducted to show the effect of low level laser therapy 810 nm and pelvic stabilization exercises has Effect on pelvic girdle pain Postpartum Pelvic girdle pain (PPGP) is common complaint in pregnant women all over the world and it has a major impact on health and functioning as it decreases quality of life. PGP generally arises in relation with pregnancy, trauma and reactive arthritis. The onset of PGP is usually by weeks 17-19 of gestation, with a peak of incidence by weeks 24- 36. Postpartum follow-up studies have shown that 5- 27% of the women had persisting pain 1-3 months after delivery. However, it was report that 7% have remaining pain 6 years after delivery causing severe discomfort and reduced ability to work , ninety prime-gravid or multigravida postnatal women's were randomly classified into three groups, Group (A): composed of 30 patients who received low-level laser therapy and pelvic stabilization exercises for 12 sessions over six week's period by 2 sessions per week. Group (B): composed of 30 patients who low-level laser therapy only for 12 sessions over six week's period by 2 sessions per week and Group (C): composed of 30 patients who received pelvic stabilization exercises For 12 sessions over six week's period by 2 sessions per week. Pain Using Visual analogue scale, serum cortisol level, and disability using pelvic girdle questionnaire) were measured and compared at 0 and 6 weeks after the treatment in the 3 groups.

DETAILED DESCRIPTION:
Study design: This work were conducted in physical therapy department of Imbaba general Hospital and in outpatient clinic of National Institute of Laser Enhanced Sciences, Cairo University Design of the study: It is a clinical study. Eighteen women's with postpartum pelvic girdle pain was participate in this study, and were randomly into three equal groups.

Eligibility Criteria:

Female participants at least ≥18 years old. Group (A): composed of 30 patients who low level laser therapy and pelvic stabilization exercises For 12 sessions over six week's period by 2 sessions per week, Group it is the study group. (B): composed of 30 patients, who low level laser therapy only for 12 sessions, over six week's period by 2 sessions per week. Group(C) .composed of 30 women's ,who received pelvic stabilization exercises only, For 12 sessions over six week's period ,by 2 sessions per week. The ethical committee clearance and an informed consent of the subjects will be taken Subjects will have all rights to withdraw from the study at any time without any responsibility.

Inclusion criteria:

1. Ongoing sacral pain with onset during the preceding pregnancy reported on a present pain drawing.
2. Pain intensity ≥4 cm as worst during the past week on a 10 cm visual analogue scale (VAS).
3. One positive pain provocation test of either Posterior Pelvic Pain Provocation test, Patrick's Faber test.
4. Provoked pain by a gentle pressure on the ischial spine, ipsilateral to reported sacral pain, at least unilaterally.

Exclusion criteria: The criteria for excluding potential research subjects included:

1. Nerve root affection in the lumbo-sacral spine
2. Inflammatory disease with pelvic bone and/or spinal manifestation
3. Known endometriosis, gynecologic cancer or ongoing malign disease.
4. Previous surgery of the lumbar spine.
5. Incapacity to complete the questionnaires.
6. Age <18 years.
7. Body mass index ≥35 kg/m2.
8. Intolerance to the treatment dose or negative reactions of the laser treatment.
9. A new pregnancy, during treatment or between the follow-ups. Study methods Instrumentation

Low-Level Laser Therapy (LLLT) parameter:

Laser medium: Semiconductor - Gallium Aluminum- Arsenide (Ga Al As). Model & manufacture: Sundom Laser-(Taiwan) RG - 300IB. Wavelength: 810 nm. Output power: 500 mw±20 Mode: Continuous Wave (CW) Spot diameter: ≤ 10 mm Treatment: 12 applications of LLLT will give on a twice weekly. Assessment procedures: Full medical history including age, BMI date of onset, medical history will collected and all patients will assessed before and after treatment program.

Outcome Measures: Primary Outcome Measure:

Pain intensity: By Visual analogue scale (VAS): Pain will assessed by using VAS that is a 10 mm calibrated line with zero representing no pain and10 representing worst pain. [Time Frame: Baseline to 6 weeks after treatment.] (Crichton 2001)

Secondary Outcome Measures:

Posterior pelvic pain provocation test (PPPPT): Used to determine the presence of sacroiliac dysfunction. It is used (often in post pregnant women) to distinguish between pelvic girdle pain and LBP: Time Frame: Baseline to 6 weeks after treatment.] (Gutke, Hansson et al. 2009) FABER Test (Patrick's test ( Flexion, Abduction and External Rotation. These three motions combined result in a clinical pain provocation test to find pathologies at the hip, lumbar and sacroiliac region. [Time Frame: Baseline to 6 weeks after treatment]. (Bagwell, Bauer et al. 2016) Pelvic Girdle Questionnaire The Pelvic Girdle Questionnaire (PGQ) is a condition-specific measure for women with pelvic girdle pain (PGP). The PGQ includes items relating to activity/participation and bodily symptoms and has reliability, validity, and feasibility for use in research and clinical practice. [Time Frame: Baseline to 6 weeks after treatment] (Stuge, Garratt et al. 2011)

Serum cortisol level:

Cortisol is a hormone secreted by the adrenal gland. It is the major corticosteroids. It is responsible for about 95% of all glucocorticoids activity in the body.(Pool and Axford 2001) It released into our body when we are under stress. Cortisol is high in subjects suffering from pain as compared with healthy and pain free subjects, as there is positive correction between the intensity of pain and increased plasma cortisol level. The blood sample will take for the measurement of plasma cortisol from 9 a.m. to 1 p.m. Each patient will be drawn two 5 ml blood samples from cubital vein two times: Time Frame: Baseline to 6 weeks after treatment. (Thabet, Hanfy et al. 2008) Treatment procedures: Eighteen women's were randomly classified into three groups.

Group (A): (study group) consist of 30 patients who received Low Level Laser Therapy and Pelvic stabilization exercise for 12 sessions .Two sessions per week over six week's period.

A) Class IV low-level laser therapy device (sundom300IB). The device delivers its energy by 2 wavelengths, 20% of the beam with 650 nm (nanometer) and 80% of the beam with 810 nm. Energy given will tested before the start of the study and once every 6 months, using Thor labs power meter PM100D and the photo sensor S 121 C, to make sure the device works correctly. The treatment applied to the sacral region by a standard laser probe at the top, and to the anterior pelvis. The physical therapist and the participant use safety eyewear during all treatment sessions and the treatment administration area is closed, have restricted access and no reflective surfaces. During treatment at sacral points, the standard probe moved 1 cm/second from a starting point to an end-point repeatedly during treatment time, bilaterally. Fluency of irradiation of 10 J/cm2, exposure of 100 seconds per point, 6 points of irradiation on the pelvic area the standard probe held perpendicular to the body surface and pressed to the skin. (Monticone, Barbarino et al. 2004) B) Pelvic stablisation exercises as in-group (C). Group (B) consist of 30 patients who received Low Level Laser Therapy only for 12 sessions .Two sessions per week over six week's period.

Group (C): (control group) consist of 30 patients will receive treatment special program of pelvic stabilization exercises only Two sessions per week over six week's period. pelvic stabilizing exercise will done by all patients in the group (C): depending on exercising of transverse abdominal in addition to co activation of lumbar multifidus muscles at the lumbosacral area ., exercising of oblique abdominal, gluteus Maximus, latissimus dorsi muscles, quadratus lumborum, erector spinae, also, hip abductors and adductors. (Mukkannavar 2013).The stress was on exercising of transverse abdominal muscles, in form of bridging exercise, posterior pelvic rocking exercise, bilateral hip abduction and adduction exercise, hip shrugging, and bilateral knees elevation. The patient lying on the side, kneeling, four points, sitting, and standing. The subjects were encouraged to activate the transversely oriented abdominal muscles regularly during daily activities. They performed two sets of exercise from 10-15 times (firstly 10 times in the 12 sessions after that15 times, for the others 12 sessions). Rest for 30-second to one minute between each set. Home program session performed for 10 minutes twice a day. Each session lasted 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Ongoing sacral pain with onset during the preceding pregnancy reported on a present pain drawing
2. Pain intensity ≥4 cm as worst during the past week on a 10 cm visual analogue scale (VAS)
3. One positive pain provocation test of either Posterior Pelvic Pain Provocation test, Patrick's Faber test.
4. Provoked pain by a gentle pressure on the ischial spine, ipsilateral to reported sacral pain, at least unilaterally.

Exclusion Criteria:

1. Nerve root affection in the lumbo-sacral spine
2. Inflammatory disease with pelvic bone and/or spinal manifestation
3. Known endometriosis, gynecologic cancer or ongoing malign disease.
4. Previous surgery of the lumbar spine.
5. Incapacity to complete the questionnaires.
6. Age <18 years.
7. Body mass index ≥35 kg/m2.
8. Intolerance to the treatment dose or negative reactions of the laser treatment.
9. A new pregnancy, during treatment or between the follow-ups. -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants at least 18 years old
Enrollment: 90 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity: | Baseline to 6 weeks after treatment .
  Pain will assessed by using VAS that is a 10 mm calibrated line with zero representing no pain and10 representing worst pain using Visual analogue scale"VAS" that is a 10 mm calibrated line with zero representing no pain and 10 representing worst pain.Worst during the past week Change from baseline to follow-up
Pelvic Girdle Questionnaire | Baseline to 6 weeks after treatment
  The Pelvic Girdle Questionnaire (PG Q) is a condition-specific measure for women with pelvic girdle pain (PGP). The questionnaire has 25 items under two sub-scales (20 items for activates and 5 items for symptoms), with percentage scores that range from 0 (no disability) to 100 (great disability),thus supplying a gap in research and clinical practice. The PG Q includes items relating to activity/participation and bodily symptoms and has reliability, validity, and feasibility for use in research and clinical practice.
Serum cortisol level: | Baseline to 6 weeks after treatment
  Cortisol is a hormone secreted by the adrenal gland. It is the major corticosteroids. It is responsible for about 95% of all glucocorticoids activity in the body.(Pool and Axford 2001) It released into our body when we are under stress. Cortisol is high in subjects suffering from pain as compared with healthy and pain free subjects, as there is positive correction between the intensity of pain and increased plasma cortisol level. The blood sample will take for the measurement of plasma cortisol from 9 a.m. to 1 p.m. Each patient will be drawn two 5 ml blood samples from cubital vein two time

SECONDARY OUTCOMES:
FABER Test (Patrick's test) | Baseline to 6 weeks after treatment
  Flexion, Abduction and External Rotation. These three motions combined result in a clinical pain provocation test to find pathologies at the hip, lumbar and sacroiliac region.
Posterior pelvic pain provocation test (PPPPT) | Baseline to 6 weeks after treatment .
  used to determine the presence of sacroiliac dysfunction. It is used (often in post pregnant women) to distinguish between pelvic girdle pain and low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Adly A Sabbour, professor, Study Director — Cairo University; Mona I Morsy, professor, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Cairo university, Giza, Cairo Governorate
  - Cairo university, Giza

IPD SHARING:
Plan to Share IPD: Yes
Methods: ninety prime-gravida or multigravida postnatal women's randomly classified into three groups, Group (A): composed of 30 patients who received pelvic stabilization exercises For 12 sessions over six week's period by 2 sessions per week. Group (B): composed of 30 patients who low-level laser therapy only for 12 sessions over six week's period by 2 sessions per week and Group(C): composed of 30 women's who received low-level laser therapy and pelvic stabilization exercises for 12 sessions over six week's period by 2 sessions per week. Pain Using Visual analogue scale, serum cortisol level, Faber test, PPPPT, and disability using pelvic girdle questionnaire were measured and compared at 0 and 6 weeks after the treatment in the 3 groups.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: started on October 2018
Access Criteria: Purpose: Postpartum Pelvic girdle pain (PPGP) is common complaint in pregnant women all over the world and it has a major impact on health and functioning as it decreases quality of life. PGP generally arises in relation with pregnancy, trauma and reactive arthritis. The onset of PGP is usually by weeks 17-19 of gestation, with a peak of incidence by weeks 24- 36. Postpartum follow-up studies have shown that 5- 27% of the women had persisting pain 1-3 months after delivery. However, it was report that 7% have remaining pain 6 years after delivery causing severe discomfort and reduced ability to work
URL: http://dr_saad2007@yahoo.com